CLINICAL TRIAL: NCT01342523
Title: Evaluation of NCI Smoking Intervention Resources
Brief Title: Evaluation of National Cancer Institute (NCI) Smoking Intervention Resources
Acronym: NCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-0007
Record Dates: First submitted 2011-03-08; First posted 2011-04-27 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Smoking Cessation; Smoking; Nicotine Dependence
Keywords: Smoking Cessation; Smoking; Nicotine
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (32):
- No CIS/No loz/No Email/Lite Website/Brief Booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, No nicotine lozenge, No motivational emails, lite website, brief mailed booklet
  Interventions: Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/No loz/No email/Lite Website/Brief booklet (Experimental): This arm of the project will address the following question:
  Does the following treatment provide efficacy relative to others:
  CIS calls, no NRT lozenge, no motivational email, Lite website, Brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- no CIS/Loz/No email/lite website/brief booklet (Experimental): This arm of the project will address the following question:
  Does this combination of services achieve effectiveness compared to others:
  No CIS phone counseling, NRT lozenge, no motivational email, lite website, brief mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- No CIS/no loz/email/lite website/brief booklet (Experimental): This arm of the project will address the following question:
  Does this combination of services lead to greater abstinence:
  No CIS counseling calls, no NRT lozenge, motivational emails, lite website, brief mailed booklet.
  Interventions: Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- No CIS/No loz/No email/Full website/Brief booklet (Experimental): This arm of the project will address the following question:
  Does this combination of services lead to greater abstinence?
  No CIS counseling, no NRT lozenge, no motivational email, full website, brief mailed booklet
  Interventions: Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- No CIS/No loz/No email/lite website/full booklet (Experimental): This arm seeks to answer the question:
  Does this combination of services achieve efficacy compared to others:
  No CIS counseling, no NRT lozenge, no motivational email, lite website, full mailed booklet
  Interventions: Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/Loz/No email/Lite website/Brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, No motivational emails, lite website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/No loz/Emails/Lite Website/Brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, No nicotine lozenge, motivational emails, lite website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/No loz/no email/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, No nicotine lozenge, No motivational emails, full website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/No loz/no email/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, No nicotine lozenge, No motivational emails, lite website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- No CIS/Loz/emails/Lite Website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, motivational emails, lite website, brief mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- No CIS/Loz/No emails/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, No motivational emails, lite website, full mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- No CIS/Loz/No emails/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, No motivational emails, full website, brief mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- no CIS/no loz/emails/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, no nicotine lozenge, motivational emails, full website, brief mailed booklet
  Interventions: Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- no CIS/no loz/emails/lite web/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, no nicotine lozenge, motivational emails, lite website, full mailed booklet
  Interventions: Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- no CIS/no loz/no email/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, no nicotine lozenge, No motivational emails, full website, full mailed booklet
  Interventions: Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/loz/emails/lite website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, motivational emails, lite website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/loz/no email/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, No motivational emails, full website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/loz/no email/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, No motivational emails, lite website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/no loz/emails/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, no nicotine lozenge, motivational emails, full website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/no loz/emails/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, no nicotine lozenge, motivational emails, lite website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/no loz/no email/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, no nicotine lozenge, No motivational emails, full website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- No CIS/loz/emails/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, motivational emails, full website, brief mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- No CIS/loz/emails/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, motivational emails, lite website, full mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- No CIS/loz/no emails/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, No motivational emails, full website, full mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- no CIS/no loz/emails/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, no nicotine lozenge, motivational emails, full website, full mailed booklet
  Interventions: Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/loz/emails/full website/brief booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, motivational emails, full website, brief mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: brief mailed booklet - smaller version of NCI's booklet
- CIS/loz/emails/lite website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, motivational emails, lite website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Lite website - lite version of smokefree.gov; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- No CIS/loz/emails/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  No CIS calls, nicotine lozenge, motivational emails, full website, full mailed booklet
  Interventions: Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/no loz/emails/full website/full booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, no nicotine lozenge, motivational emails, full website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/Loz/no Emails/Full Website/Full Booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, No motivational emails, full website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide
- CIS/Loz/Emails/Full Website/Full Booklet (Experimental): This arm of the project will address the following question:
  How effective is the following intervention?
  CIS calls, nicotine lozenge, motivational emails, full website, full mailed booklet
  Interventions: Other: CIS - telephone cessation quitline counseling; Other: Lozenge - nicotine mini-lozenges; Other: Emails - Brief smoking prevention messages; Other: Full website - standard smokefree.gov website content; Other: Full mailed booklet - NCI's detailed 36-page quit guide

INTERVENTIONS:
Other: CIS - telephone cessation quitline counseling — Up to 5 total tobacco cessation counseling calls
  Arms: CIS/Loz/Emails/Full Website/Full Booklet; CIS/Loz/No email/Lite website/Brief booklet; CIS/Loz/no Emails/Full Website/Full Booklet; CIS/No loz/Emails/Lite Website/Brief booklet; CIS/No loz/No email/Lite Website/Brief booklet; CIS/No loz/no email/full website/brief booklet; CIS/No loz/no email/lite website/full booklet; CIS/loz/emails/full website/brief booklet; CIS/loz/emails/lite website/brief booklet; CIS/loz/emails/lite website/full booklet; CIS/loz/no email/full website/brief booklet; CIS/loz/no email/lite website/full booklet; CIS/no loz/emails/full website/brief booklet; CIS/no loz/emails/full website/full booklet; CIS/no loz/emails/lite website/full booklet; CIS/no loz/no email/full website/full booklet
Other: Lozenge - nicotine mini-lozenges — 2-week starter pack of nicotine mini-lozenges
  Arms: CIS/Loz/Emails/Full Website/Full Booklet; CIS/Loz/No email/Lite website/Brief booklet; CIS/Loz/no Emails/Full Website/Full Booklet; CIS/loz/emails/full website/brief booklet; CIS/loz/emails/lite website/brief booklet; CIS/loz/emails/lite website/full booklet; CIS/loz/no email/full website/brief booklet; CIS/loz/no email/lite website/full booklet; No CIS/Loz/No emails/full website/brief booklet; No CIS/Loz/No emails/lite website/full booklet; No CIS/Loz/emails/Lite Website/brief booklet; No CIS/loz/emails/full website/brief booklet; No CIS/loz/emails/full website/full booklet; No CIS/loz/emails/lite website/full booklet; No CIS/loz/no emails/full website/full booklet; no CIS/Loz/No email/lite website/brief booklet
Other: Emails - Brief smoking prevention messages — Brief email messages that could be accessed by any computer or mobile device that allowed email receipt
  Arms: CIS/Loz/Emails/Full Website/Full Booklet; CIS/No loz/Emails/Lite Website/Brief booklet; CIS/loz/emails/full website/brief booklet; CIS/loz/emails/lite website/brief booklet; CIS/loz/emails/lite website/full booklet; CIS/no loz/emails/full website/brief booklet; CIS/no loz/emails/full website/full booklet; CIS/no loz/emails/lite website/full booklet; No CIS/Loz/emails/Lite Website/brief booklet; No CIS/loz/emails/full website/brief booklet; No CIS/loz/emails/full website/full booklet; No CIS/loz/emails/lite website/full booklet; No CIS/no loz/email/lite website/brief booklet; no CIS/no loz/emails/full website/brief booklet; no CIS/no loz/emails/full website/full booklet; no CIS/no loz/emails/lite web/full booklet
Other: Full website - standard smokefree.gov website content — Over 50 web pages of resources for quitting smoking, including interactive features and referral links
  Arms: CIS/Loz/Emails/Full Website/Full Booklet; CIS/Loz/no Emails/Full Website/Full Booklet; CIS/No loz/no email/full website/brief booklet; CIS/loz/emails/full website/brief booklet; CIS/loz/no email/full website/brief booklet; CIS/no loz/emails/full website/brief booklet; CIS/no loz/emails/full website/full booklet; CIS/no loz/no email/full website/full booklet; No CIS/Loz/No emails/full website/brief booklet; No CIS/No loz/No email/Full website/Brief booklet; No CIS/loz/emails/full website/brief booklet; No CIS/loz/emails/full website/full booklet; No CIS/loz/no emails/full website/full booklet; no CIS/no loz/emails/full website/brief booklet; no CIS/no loz/emails/full website/full booklet; no CIS/no loz/no email/full website/full booklet
Other: Lite website - lite version of smokefree.gov — Reduced version of the smokefree.gov website developed for the research; reduced number of web pages and external links (considered a placebo intervention)
  Arms: CIS/Loz/No email/Lite website/Brief booklet; CIS/No loz/Emails/Lite Website/Brief booklet; CIS/No loz/No email/Lite Website/Brief booklet; CIS/No loz/no email/lite website/full booklet; CIS/loz/emails/lite website/brief booklet; CIS/loz/emails/lite website/full booklet; CIS/loz/no email/lite website/full booklet; CIS/no loz/emails/lite website/full booklet; No CIS/Loz/No emails/lite website/full booklet; No CIS/Loz/emails/Lite Website/brief booklet; No CIS/No loz/No Email/Lite Website/Brief Booklet; No CIS/No loz/No email/lite website/full booklet; No CIS/loz/emails/lite website/full booklet; No CIS/no loz/email/lite website/brief booklet; no CIS/Loz/No email/lite website/brief booklet; no CIS/no loz/emails/lite web/full booklet
Other: Full mailed booklet - NCI's detailed 36-page quit guide — NCI's Clearing the Air brochure for preparing to quit, quitting and preventing relapse
  Arms: CIS/Loz/Emails/Full Website/Full Booklet; CIS/Loz/no Emails/Full Website/Full Booklet; CIS/No loz/no email/lite website/full booklet; CIS/loz/emails/lite website/full booklet; CIS/loz/no email/lite website/full booklet; CIS/no loz/emails/full website/full booklet; CIS/no loz/emails/lite website/full booklet; CIS/no loz/no email/full website/full booklet; No CIS/Loz/No emails/lite website/full booklet; No CIS/No loz/No email/lite website/full booklet; No CIS/loz/emails/full website/full booklet; No CIS/loz/emails/lite website/full booklet; No CIS/loz/no emails/full website/full booklet; no CIS/no loz/emails/full website/full booklet; no CIS/no loz/emails/lite web/full booklet; no CIS/no loz/no email/full website/full booklet
Other: brief mailed booklet - smaller version of NCI's booklet — 12-page booklet developed by the investigators for the research (considered to be placebo intervention)
  Arms: CIS/Loz/No email/Lite website/Brief booklet; CIS/No loz/Emails/Lite Website/Brief booklet; CIS/No loz/No email/Lite Website/Brief booklet; CIS/No loz/no email/full website/brief booklet; CIS/loz/emails/full website/brief booklet; CIS/loz/emails/lite website/brief booklet; CIS/loz/no email/full website/brief booklet; CIS/no loz/emails/full website/brief booklet; No CIS/Loz/No emails/full website/brief booklet; No CIS/Loz/emails/Lite Website/brief booklet; No CIS/No loz/No Email/Lite Website/Brief Booklet; No CIS/No loz/No email/Full website/Brief booklet; No CIS/loz/emails/full website/brief booklet; No CIS/no loz/email/lite website/brief booklet; no CIS/Loz/No email/lite website/brief booklet; no CIS/no loz/emails/full website/brief booklet

SUMMARY:
This is an evaluative study of three National Cancer Institute (NCI) smoking cessation resources: specifically, the smokefree.gov and women smokefree.gov websites, and the CIS counseling phone calls. The following are the identified critical questions: (1). How effective is each of the tobacco interventions (websites [smokefree.gov & women smokefree.gov], NCI's Cessation Quitline counseling services operated by the Cancer Information Service (CIS) (2). How do they compare with alternative intervention strategies? (3). Which types of interventions appear to work best together (due to additive or interactive effects)? (4). How do these interventions work? (5). How much are these interventions used, and what are their relative use rates? (6). Are there important differences in effectiveness or use rates as a function of gender, SES, or other important person factors? We believe that the research study will address all of these questions, as well as some less central ones.

DETAILED DESCRIPTION:
This an evaluative study of three National Cancer Institute (NCI) smoking cessation resources: specifically, the smokefree.gov and women smokefree.gov websites, and the CIS counseling phone calls. The following are the identified critical questions: (1). How effective is each of the tobacco interventions (websites [smokefree.gov & women smokefree.gov], NCI's Cessation Quitline counseling services operated by the Cancer Information Service (CIS) (2). How do they compare with alternative intervention strategies? (3). Which types of interventions appear to work best together (due to additive or interactive effects)? (4). How do these interventions work? (5). How much are these interventions used, and what are their relative use rates? (6). Are there important differences in effectiveness or use rates as a function of gender, SES, or other important person factors? We believe that the research study will address all of these questions, as well as some less central ones.

The primary goal of this research is to obtain experimental data on the effectiveness of the major eHealth and communication smoking cessation interventions (smokefree.gov, women smokefree.gov, and NCI's Quitline counseling services). The primary bases for comparison would be quit attempts and cessation success, and each intervention would be compared with a control condition not receiving the intervention. In addition to the targeted interventions, participants may also be assigned to several different comparison interventions: i.e., email prompts, mailings/brochures, and OTC nicotine medication. The resulting data would allow us to determine effect sizes for each type of intervention relative to a control condition, which would allow us to determine the relative effectiveness of each intervention: i.e., how well the interventions stack-up against one another in terms of effect sizes.

Secondary goals of this research are to:

1. . Determine how much the participants use the interventions;
2. . Determine the mechanisms of benefit (perform meditational analyses);
3. . Compare benefits for important smoker populations;
4. . Determine whether any of the interventions produce subtractive or synergistic effects; and
5. . Obtain basic health economic estimates such as cost/quitter.

The project will also include a substudy directed toward pregnant women and women who are interested in participating but are unwilling to agree to utilize approved contraceptive methods for the duration of the study. This substudy will utilize all of the treatment conditions except the medication condition, since medication is not recommended for women who are pregnant in the US. Department of Health and Human Services treatment guideline for tobacco dependence

ELIGIBILITY:
Inclusion Criteria:

(1). Interest in quitting smoking within the next 30 days, but not already actively engaged in quitting (e.g., subject should not be currently participating in other cessation counseling or taking cessation medication treatment for the purpose of a quit attempt); (2). The person has a phone and has home internet access; (3). The person has an email address that can be used to send assessments, and deliver email prompts; (4). The person expresses willingness to provide assessment information and have his/her computer use of the assigned website tracked; (5). There are contraindications to over the counter nicotine replacement therapy (NRT) use (e.g., pregnancy); (6). The person smokes ≥ 5 cpd; (7). The person is ≥ 18 years;(8). The person accesses the internet with no more than 3 computers/devices (including devices such as iPads and smartphones); and (9). No other members of the person's household are participating in the NCI website evaluation. (The age restriction is due to the possible assignment to medication, which is not recommended for adolescents.) Subjects will not have to express an interest in using NRT. They may be sent NRT depending upon experimental assignment, but a commitment to use medication is not a requirement of participation. Also, pregnant smokers, or those who believe they may become pregnant, can participate, but they will be randomly assigned to only the non-medication treatments and participate only in the substudy. [They will not be included in the regular data analyses, and power will be too small to permit meaningful inferential tests. However, effect sizes in this small group of smokers will be determined for comparison with the effect sizes obtained in the main study.] Due to limitations in the volume of new calls that can be handled in the phone counseling component, recruitment will not exceed 300 per month. When monthly recruitment goal has been met, the recruitment invitation will be turned off until the following month. At the point where it is necessary to achieve the desired (50/50) gender balance, the invitation to participate in the study will be restricted by sex until full enrollment is achieved.

Exclusion Criteria:

(1). If the person has no interest in quitting smoking within the next 30 days or if the person is actively engaged in quitting (e.g., subject is currently participating in other cessation counseling or taking cessation medication treatment for the purpose of a quit attempt); (2). Person does not have a phone or home internet access; (3). The person does not have an email address that can be used to send assessments, and deliver email prompts; (4). The person is not willing to provide assessment information and have his/her computer use of the assigned website tracked; (5). There are contraindications to over the counter nicotine replacement therapy (NRT) use (e.g., pregnancy); (6). The person smokes < 5 cpd; (7). The person is <18 years;(8). The person accesses the internet with more than 4 computers (including devices such as iPads and smartphones); and (9). One or more members of the person's household are already participating in the NCI website evaluation. (The age restriction is due to the possible assignment to medication, which is not recommended for adolescents.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/
- See also: Smokefree.gov — http://www.smokefree.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period ran from November 28, 2011 through March 26, 2013. All study participants were recruited through the portal to the smokefree.gov website.
Pre-assignment Details: Prior to randomization, potential participants were asked to make a "confirmation" call to an automated answering system to confirm willingness to perform study procedures. The call was intended to increase the likelihood that individuals would take treatment and follow-up calls. Randomization occurred immediately after the confirmation call.
Period: Overall Study
Arm/Group | No CIS/No Loz/No Email/Lite Website/Brief Booklet | CIS/No Loz/No Email/Lite Website/Brief Booklet | no CIS/Loz/No Email/Lite Website/Brief Booklet | No CIS/no Loz/Email/Lite Website/Brief Booklet | No CIS/No Loz/No Email/Full Website/Brief Booklet | No CIS/No Loz/No Email/Lite Website/Full Booklet | CIS/Loz/No Email/Lite Website/Brief Booklet | CIS/No Loz/Emails/Lite Website/Brief Booklet | CIS/No Loz/no Email/Full Website/Brief Booklet | CIS/No Loz/no Email/Lite Website/Full Booklet | No CIS/Loz/Emails/Lite Website/Brief Booklet | No CIS/Loz/No Emails/Lite Website/Full Booklet | No CIS/Loz/No Emails/Full Website/Lite Booklet | no CIS/no Loz/Emails/Full Website/Brief Booklet | no CIS/no Loz/Emails/Lite Web/Full Booklet | no CIS/no Loz/no Email/Full Website/Full Booklet | CIS/Loz/Emails/Lite Website/Brief Booklet | CIS/Loz/no Email/Full Website/Brief Booklet | CIS/Loz/no Email/Lite Website/Full Booklet | CIS/no Loz/Emails/Full Website/Brief Booklet | CIS/no Loz/Emails/Lite Website/Full Booklet | CIS/no Loz/no Email/Full Website/Full Booklet | No CIS/Loz/Emails/Full Website/Brief Booklet | No CIS/Loz/Emails/Lite Website/Full Booklet | No CIS/Loz/no Emails/Full Website/Full Booklet | no CIS/no Loz/Emails/Full Website/Full Booklet | CIS/Loz/Emails/Full Website/Brief Booklet | CIS/Loz/Emails/Lite Website/Full Booklet | No CIS/Loz/Emails/Full Website/Full Booklet | CIS/no Loz/Emails/Full Website/Full Booklet | CIS/Loz/no Emails/Full Website/Full Booklet | CIS/Loz/Emails/Full Website/Full Booklet
Started | 35 | 32 | 36 | 33 | 36 | 36 | 22 | 27 | 28 | 28 | 38 | 38 | 39 | 38 | 38 | 32 | 29 | 27 | 21 | 27 | 29 | 30 | 36 | 36 | 37 | 38 | 34 | 31 | 35 | 29 | 31 | 28
Completed | 34 | 32 | 36 | 32 | 36 | 36 | 22 | 27 | 28 | 28 | 38 | 36 | 39 | 36 | 37 | 32 | 28 | 27 | 21 | 27 | 29 | 30 | 36 | 35 | 36 | 36 | 33 | 30 | 34 | 28 | 30 | 27
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No CIS/No Loz/No Email/Lite Website/Brief Booklet | CIS/No Loz/No Email/Lite Website/Brief Booklet | no CIS/Loz/No Email/Lite Website/Brief Booklet | No CIS/no Loz/Email/Lite Website/Brief Booklet | No CIS/No Loz/No Email/Full Website/Brief Booklet | No CIS/No Loz/No Email/Lite Website/Full Booklet | CIS/Loz/No Email/Lite Website/Brief Booklet | CIS/No Loz/Emails/Lite Website/Brief Booklet | CIS/No Loz/no Email/Full Website/Brief Booklet | CIS/No Loz/no Email/Lite Website/Full Booklet | No CIS/Loz/Emails/Lite Website/Brief Booklet | No CIS/Loz/No Emails/Lite Website/Full Booklet | No CIS/Loz/No Emails/Full Website/Lite Booklet | no CIS/no Loz/Emails/Full Website/Brief Booklet | no CIS/no Loz/Emails/Lite Web/Full Booklet | no CIS/no Loz/no Email/Full Website/Full Booklet | CIS/Loz/Emails/Lite Website/Brief Booklet | CIS/Loz/no Email/Full Website/Brief Booklet | CIS/Loz/no Email/Lite Website/Full Booklet | CIS/no Loz/Emails/Full Website/Brief Booklet | CIS/no Loz/Emails/Lite Website/Full Booklet | CIS/no Loz/no Email/Full Website/Full Booklet | No CIS/Loz/Emails/Full Website/Brief Booklet | No CIS/Loz/Emails/Lite Website/Full Booklet | No CIS/Loz/no Emails/Full Website/Full Booklet | no CIS/no Loz/Emails/Full Website/Full Booklet | CIS/Loz/Emails/Full Website/Brief Booklet | CIS/Loz/Emails/Lite Website/Full Booklet | No CIS/Loz/Emails/Full Website/Full Booklet | CIS/no Loz/Emails/Full Website/Full Booklet | CIS/Loz/no Emails/Full Website/Full Booklet | CIS/Loz/Emails/Full Website/Full Booklet | Total
Number analyzed (Participants) | 35 | 32 | 36 | 33 | 36 | 36 | 22 | 27 | 28 | 28 | 38 | 38 | 39 | 38 | 38 | 32 | 29 | 27 | 21 | 27 | 29 | 30 | 36 | 36 | 37 | 38 | 34 | 31 | 35 | 29 | 31 | 28 | 1034
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5
  Between 18 and 65 years | 34 | 32 | 35 | 32 | 36 | 36 | 22 | 26 | 27 | 28 | 38 | 38 | 37 | 37 | 37 | 32 | 28 | 25 | 21 | 27 | 29 | 27 | 36 | 35 | 35 | 37 | 33 | 29 | 35 | 28 | 29 | 27 | 1008
  >=65 years | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.117) | 41.97 (12.124) | 39.47 (11.661) | 40.58 (13.709) | 39.89 (12.132) | 39.92 (13) | 40.5 (11.859) | 38.52 (14.091) | 37.71 (13.160) | 38.11 (13.076) | 39 (12.192) | 39.16 (10.812) | 36.03 (11.957) | 39.47 (12.967) | 38.18 (11.925) | 40.56 (11.007) | 42.31 (13.134) | 43.04 (12.738) | 35.76 (12.373) | 39.26 (10.376) | 37.79 (10.115) | 40.37 (13.433) | 38.81 (11.112) | 42.97 (13.716) | 38.92 (13.215) | 40.32 (11.242) | 38.47 (12.310) | 37.77 (13.386) | 36.91 (10.441) | 35.62 (12.754) | 38.23 (13.674) | 42.54 (12.96) | 39.28 (12.343)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 27 | 23 | 21 | 23 | 19 | 19 | 19 | 23 | 24 | 25 | 25 | 21 | 26 | 23 | 23 | 21 | 13 | 19 | 17 | 19 | 23 | 28 | 28 | 25 | 18 | 24 | 22 | 20 | 25 | 22 | 703
  Male | 15 | 14 | 9 | 10 | 15 | 13 | 3 | 8 | 9 | 5 | 14 | 13 | 14 | 17 | 12 | 9 | 6 | 6 | 8 | 8 | 12 | 11 | 13 | 8 | 9 | 13 | 16 | 7 | 13 | 9 | 6 | 6 | 331
Region of Enrollment [Number; unit: participants]
  United States | 35 | 32 | 36 | 33 | 36 | 36 | 22 | 27 | 28 | 28 | 38 | 38 | 39 | 38 | 38 | 32 | 29 | 27 | 21 | 27 | 29 | 30 | 36 | 36 | 37 | 38 | 34 | 31 | 35 | 29 | 31 | 28 | 1034

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point-Prevalence Abstinence From Smoking
Description: Abstinence will be defined as 7-day point prevalence.
Time Frame: Measured after the 3 month follow up assessment
Population: "Intention to treat (ITT)
Measure: Number; unit: percentage of participants not smoking
Groups:
- Cancer Information Service Counseling ("CIS"): Participants in this intervention group received telephone quitline counseling from the Cancer Information Service (CIS). These proactive calls initiated by CIS included an initial call (30 min), occurring within 3 days of enrollment, plus 4 additional counseling calls (up to 15 min each) scheduled to occur on the quit day or the day after, and then weekly for the next 3 weeks. The content of the counseling calls focused initially on motivating quitting and then setting a quit date, providing support, building self-efficacy, and skill training. The CIS intervention group will be compared to a "No CIS" group. The original randomization plan called for approximately half of the total sample of 1034 participants to be randomized to this intervention group (CIS) and the other half to the No CIS intervention group. However, due to a problem in the electronic transfer of data from the research coordinating site to CIS, 453 participants were randomized to CIS and 581 to the "No CIS" group.
- No Cancer Information Service Counseling ("No CIS"): Participants in this intervention group did not receive telephone quitline counseling from the Cancer Information Service (CIS). This intervention group will be compared to an intervention group that did receive telephone quitline counseling from the CIS. The original randomization plan called for approximately half of the total sample of 1034 participants to be randomized to this intervention group (No CIS) and the other half to the CIS intervention group. However, due to a problem in the electronic transfer of data from the research coordinating site to CIS, 581 participants were randomized to "No CIS" group and 453 to the CIS group.
- Nicotine Replacement Therapy (NRT; Mini-Lozenge for 2 Weeks): Participants in this intervention group received a 2-week starter package of nicotine mini-lozenges, with dose based on time to since first cigarette of the day as per package instructions. Each package contained 2 mini-lozenge dispensers (162 lozenges total) and instructions on proper use. Approximately half of the total sample of 1034 participants was randomized to receive the 2-week supply of mini-lozenges; the other half received no mini-lozenges.
- No Nicotine Replacement Therapy: Participants in this intervention group received no nicotine replacement therapy (NRT), i.e., no nicotine mini-lozenges. Approximately half of the total sample of 1034 participants was randomized to receive no NRT; the other half a 2-week supply of nicotine mini-lozenges.
- Email Messaging: Participants Email Messaging intervention group received brief email messages that could be accessed by any computer or mobile device that allowed email receipt. Messages were intended to provide: (1) Motivation/encouragement; (2) Quitting tips and information; (3) Adherence/education prompts (to use available resources as recommended), and (4) relapse prevention content. These emailed messages were sent twice/day for two weeks, once/day for an additional month, and then one every 3rd day for an additional 6 weeks (constituting a 3-month-long intervention). Approximately half of the total sample of 1034 participants was randomized to receive Email Messaging; the other half received no Email Messaging.
- No Email Messaging: Participants in this intervention group received no Email Messaging. Approximately half of the total sample of 1034 participants was randomized to receive no Email Messaging; the other half received 3 months of Email Messaging.
- Full SmokeFree.Gov Website: Participants in the Full SmokeFree.gov website intervention group received the standard smokefree.gov website content that included resources to motivate quitting and a step-by-step quitting guide that provided a skill-based intervention for preparing to quit, quitting, and maintaining abstinence. In addition, the active website offered encouragement and support, motivational information, and interactive features and referral links. The active website did not include direct interaction with users (e.g. live help) or interactive audio or video content. User-engagement features included task charts for behavior change, self-monitoring tools (e.g. for cravings and self-assessment), creation of a personal calendar, links to a quitline or to a counselor via text message for live help and social support through social media. No tailoring, feedback or outbound reminders were in use. Approximately half of the total sample of 1034 participants was randomized to receive the Full Smoke
- Lite SmokeFree.Gov Website: Participants in the Lite SmokeFree.gov Website intervention group received received the "Lite" version of the website (developed by the investigators for this research) that included information about smoking and health such as benefits of quitting and information about withdrawal, medications and stress, but contained no interactive features or content that would support skill training. The look and graphics directly mirrored the full smokefree.gov website, but the number of web pages was reduced from over 50 to 16, and external links to resources were virtually eliminated. Approximately half of the total sample of 1034 participants was randomized to receive theLite SmokeFree.gov Website; the other half received the Full SmokeFree.gov Website.
- Full Cessation Booklet: Participants in the Full Cessation Booklet intervention group received the National Cancer Institute's 36-page "Clearing the Air" brochure (www.smokefree.gov/pubs/clearing_the_air.pdf), containing a detailed guide for preparing to quit, quitting, and preventing relapse as well as suggested resources. Approximately half of the total sample of 1034 participants was randomized to receive the Full Cessation Booklet; the other half received a Brief Cessation Booklet.
- Brief Cessation Booklet: Participants in the Full Cessation Booklet intervention group received a 12-page booklet developed by the investigators. The content of this booklet was the same as contained in the 36-page "Clearing the Air" booklet except that information directly relevant to coping skill training (identification of smoking triggers, making coping plans) was removed. Approximately half of the total sample of 1034 participants was randomized to receive the Brief Cessation Booklet; the other half received the Full Cessation Booklet.
Arm/Group | Cancer Information Service Counseling ("CIS") | No Cancer Information Service Counseling ("No CIS") | Nicotine Replacement Therapy (NRT; Mini-Lozenge for 2 Weeks) | No Nicotine Replacement Therapy | Email Messaging | No Email Messaging | Full SmokeFree.Gov Website | Lite SmokeFree.Gov Website | Full Cessation Booklet | Brief Cessation Booklet
Number analyzed (Participants) | 453 | 581 | 518 | 516 | 526 | 508 | 525 | 509 | 517 | 517
percentage of participants not smoking | 27.8 | 26.3 | 30.5 | 23.4 | 26.2 | 27.8 | 29.5 | 24.4 | 26.3 | 27.7
Statistical Analysis 1: Comparison: Cancer Information Service Counseling ("CIS") vs No Cancer Information Service Counseling ("No CIS"); Null hypothesis: No difference in 3-month abstinence rates for participants receiving CIS vs No CIS. We hypothesized that CIS would result in significantly higher abstinence rates compared to No CIS; Test type: Superiority or Other; p = .825, Regression, Logistic — P-value is not adjusted for multiple comparisons; The logistic regression model included all 5 treatment main effects and the 10 two-way interactions as well as gender, race, and age as covariates; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.88 to 1.17]
Statistical Analysis 2: Comparison: Nicotine Replacement Therapy (NRT; Mini-Lozenge for 2 Weeks) vs No Nicotine Replacement Therapy; Null hypothesis: No difference in 3-month abstinence rates for participants receiving NRT vs No NRT. We hypothesized that NRT would result in significantly higher abstinence rates compared to No NRT; Test type: Superiority or Other; p = .028, Regression, Logistic — P-value is not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [1.02 to 1.36]
Statistical Analysis 3: Comparison: Email Messaging vs No Email Messaging; Null hypothesis: No difference in 3-month abstinence rates for participants receiving Email Messaging vs No Email Messaging. We hypothesized that Email Messaging would result in significantly higher abstinence rates compared to No Email Messaging; Test type: Superiority or Other; p = .755, Regression, Logistic — P-value is not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.85 to 1.13]
Statistical Analysis 4: Comparison: Full SmokeFree.Gov Website vs Lite SmokeFree.Gov Website; Null hypothesis: No difference in 3-month abstinence rates for participants receiving the Full SmokeFree.gov Website vs the Lite SmokeFree.gov Website . We hypothesized that the Full SmokeFree.gov Website would result in significantly higher abstinence rates compared to the LiteSmokeFree.gov Website; Test type: Superiority or Other; p = .057, Regression, Logistic — P-value is not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.996 to 1.33]
Statistical Analysis 5: Comparison: Full Cessation Booklet vs Brief Cessation Booklet; Null hypothesis: No difference in 3-month abstinence rates for participants receiving the Full Cessation Booklet vs the Brief Cessation Booklet We hypothesized that the Full Cessation Booklet would result in significantly higher abstinence rates compared to the Brief Cessation Booklet; Test type: Superiority or Other; p = .555, Regression, Logistic — P-value is not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI [0.83 to 1.11]

2. Secondary Outcome: Smoking Outcomes
Description: Inclusive of smoking rate amongst those smoking, smoking cessation milestones: initial cessation, lapse latency, lapse-relapse latency; and setting a quit date.
Time Frame: Measured at the1 week, 2 week, 3 week, 1 month, 3 month and 7 month follow up assessments.
Reporting Status: Not Posted

3. Secondary Outcome: Resource Use/Engagement
Description: We will measure participants' use the experimental resources compared to the non-experimental resources. Particularly with the study websites, we will be tracking how often and how long participants use the regular smokefree.gov website versus the placebo website as well as what parts of the websites they are using for 6 months.
Time Frame: Assessed at the 7 month follow up assessment. Furthermore, Website use will be collected as pages viewed, time viewed, use occasions, and composite measures. Counseling use will be measured by number of counseling calls.
Reporting Status: Not Posted

4. Secondary Outcome: Effectiveness of the Experimental Resources.
Description: We will measure how these experimental resources (as well as combinations of resources) aid in quit attempts and abstinence outcomes.
Time Frame: Data collected at all assessments (Measured at the1 week, 2 week, 3 week, 1 month, 3 month and 7 month follow ups), during web use measurements (6 months), and counseling calls measurements (4 weeks). Analyzed after the study.
Reporting Status: Not Posted

5. Secondary Outcome: Withdrawal Symptoms
Description: We will measure the manifestation and severity of withdrawal symptoms of participants in each treatment group.
Time Frame: Measured at the1 week, 2 week, 3 week, 1 month, 3 month and 7 month follow up assessments.
Reporting Status: Not Posted

6. Secondary Outcome: Perceived Support
Description: We will measure perceived support from both treatment and non-treatment resources.
Time Frame: Measured at the1 month, 3 month and 7 month follow up assessments.
Reporting Status: Not Posted

7. Secondary Outcome: Treatment Satisfaction
Description: We will measure how satisfied participants were with the resources they were given as well as what might have made their quit attempts easier or more successful.
Time Frame: Measured at the 1 month, 3 month and 7 month follow up assessments
Reporting Status: Not Posted

8. Secondary Outcome: Increased Quit Attempts
Description: Quit attempts will be defined in two ways: self-report of a serious attempt to quit, and occurrence of at least a 24 hr period of abstinence that was for the purpose of cessation.
Time Frame: Measured at the 1 month, 3 month and 7 month follow up assessments.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were only collected for the lozenge condition, since no other treatments had the potential to cause an adverse event.
Groups:
- Lozenge: 2 week supply of nicotine mini-lozenge. This is the only study arm for which adverse events were appropriate to be collected and analyzed, since all other arms did not involve interventions that could generate an adverse event report.
Arm/Group | Lozenge
Serious Adverse Events (participants affected / at risk) | 0/518
Other Adverse Events (participants affected / at risk) | 0/518

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No